CLINICAL TRIAL: NCT05280769
Title: Effects of an Oral Nicotine Product in Smokeless Tobacco Users
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: HM20018418; U54DA036105 (NIH)
Record Dates: First submitted 2022-03-04; First posted 2022-03-15 (Actual); Last update posted 2024-10-02 (Actual); Status verified 2024-09

CONDITIONS: Tobacco Use
MeSH Terms: conditions — Tobacco Use | interventions — Tobacco, Smokeless

STUDY DESIGN:
Intervention Model Description: Single arm study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single arm design (Experimental): On four separate occasions, participants will come to the research center and be asked to use a nicotine pouch or smokeless tobacco provided by the study team two separate times. The nicotine pouches or smokeless tobacco contain different amounts of nicotine. Participants will not know the concentration of nicotine in the nicotine pouch, but they will know the concentration and brand of the smokeless tobacco (it will be their usual brand). All participants will complete all four study conditions.
  Interventions: Other: oral nicotine pouch - 2 mg; Other: oral nicotine pouch - 4 mg; Other: oral nicotine pouch - 8 mg; Other: Smokeless tobacco

INTERVENTIONS:
Other: oral nicotine pouch - 2 mg — "On" brand oral nicotine pouch with 2 mg of protonated nicotine in "original" flavor
Other: oral nicotine pouch - 4 mg — "On" brand oral nicotine pouch with 4 mg of protonated nicotine in "original" flavor
Other: oral nicotine pouch - 8 mg — "On" brand oral nicotine pouch with 8 mg of protonated nicotine in "original" flavor
Other: Smokeless tobacco — Participant's typical brand of smokeless tobacco

SUMMARY:
The purpose of this research study is to find out how three different nicotine pouches and participant's own brand of smokeless tobacco affect blood nicotine levels and how participants feel.

ELIGIBILITY:
Inclusion Criteria:

* Healthy (determined by self-report)
* Between the ages of 18-55
* Willing to provide informed consent, attend the lab sessions and abstain from tobacco/nicotine as required
* Agree to use designated products according to study protocol
* Smokeless tobacco users and must report using smokeless tobacco daily. Smokeless tobacco users must have a 'positive' cotinine cassette result to verify nicotine use

Exclusion Criteria:

* The following self-reported current, diagnosed medical condition(s): heart-related conditions (e.g., recent heart attack/stroke, coronary heart disease), severe immune system disorders (e.g., HIV/AIDS, multiple sclerosis), respiratory disorders (e.g., COPD, asthma), kidney diseases, liver diseases (e.g., cirrhosis), or seizures
* Other self-reported current, diagnosed medical conditions (e.g., diabetes, thyroid disease, Lyme disease) may be excluded after consultation with the PI and medical monitor: any medical condition/medication that may affect participant safety, study outcomes, or biomarker data will be excluded based on these consultations
* Self-reported current, diagnosed psychiatric conditions, and who are currently under the care of a physician for psychiatric conditions, or who report current psychiatric treatment or psychotropic medication use
* Not providing answers to questions related to inclusion/exclusion criteria
* Breast-feeding or pregnant women (pregnancy tested by urinalysis at screening
* Weigh less than 110 pounds
* Intend to quit tobacco/nicotine use in the next 30 days

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2022-08-23 (Actual); Primary Completion 2023-11-28 (Actual); Study Completion 2023-11-28 (Actual)

PRIMARY OUTCOMES:
Change in Plasma nicotine concentration | Baseline to the end of the session, approximately 4 hours
  Blood will be taken multiple times in each session to assess the extent to which product use changes plasma nicotine levels compared to baseline

OTHER OUTCOMES:
Change physical sensations | Baseline to the end of the session, approximately 4 hours
  The Direct Effects of Nicotine Questionnaire (DEN) is used to assess the extent to which product use affects participants physically. It consists of 10 items, each of which is scored from 0 - 100 with 0 being not at all and 100 being extremely.
Change in sensations and emotions | Baseline to the end of the session, approximately 4 hours
  The Direct Effects of Smokeless Tobacco (DESLT) Questionnaire is used to assess sensations and emotions associated with smokeless tobacco use. It consists of 12 items, each of which is scored from 0 - 100 with 0 being not at all and 100 being extremely.
Change emotions and urges | Baseline to the end of the session, approximately 4 hours
  The Hughes-Hatsukami Questionnaire (HH) is used to assess the extent to which product use affects a variety of emotions and urges. It consists of 11 items, each of which is scored from 0 - 100 with 0 being not at all and 100 being extremely.

CONTACTS AND LOCATIONS:
Overall Officials: Alison Breland, PhD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No